CLINICAL TRIAL: NCT00683124
Title: Effects of Losartan vs. Nebivolol vs. the Association of Both on the Progression of Aortic Root Dilation in Marfan Syndrome (MFS) With FBN1 Gene Mutations.
Brief Title: Nebivolol Versus Losartan Versus Nebivolol+Losartan Against Aortic Root Dilation in Genotyped Marfan Patients
Acronym: MaNeLo
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Menarini Group (Industry)
Responsible Party: Doctor Eloisa Arbustini, MD, FESC, FACC, IRCCS Foundation San Matteo Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FARM7KP2PX; EudraCT 2008-001462-81
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Marfan Syndrome
Keywords: Marfan Syndrome; Losartan; Nebivolol; Transforming Growth Factor Beta; Aortic Root Dilation
MeSH Terms: conditions — Marfan Syndrome; Camurati-Engelmann Syndrome | interventions — Losartan; Nebivolol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Losartan (Experimental): Losartan administered as maximal tolerated dosage, not to exceed the maximal theorical dosage of 100 mg/day for adults and 1,6 mg/kg/die for children minor than 16 years.
  Interventions: Drug: Losartan
- Nebivolol (Experimental): Nebivolol administered as maximal tolerated dosage, not to exceed the maximal theorical dosage of 10 mg/day for adults and 0,16 mg/kg/die for children minor than 16 years.
  Interventions: Drug: Nebivolol
- Losartan+Nebivolol (Experimental): Losartan administered as maximal tolerated dosage, not to exceed the maximal theorical dosage of 100 mg/day for adults and 1,6 mg/kg/die for children minor than 16 years.
  Nebivolol administered as maximal tolerated dosage, not to exceed the maximal theorical dosage of 10 mg/day for adults and 0,16 mg/kg/die for children minor than 16 years.
  Interventions: Drug: Losartan and nebivolol

INTERVENTIONS:
Drug: Losartan and nebivolol — Nebivolol is administered orally as pills. It is given preferentially once a day in the morning or, if not well tolerated because of hypotension, the total daily dosage is given in two administrations.
  Losartan is administered orally as pills. It is given preferentially once a day or, if not well tolerated because of hypotension, the total daily dosage is given in two administrations
  Arms: Losartan+Nebivolol
Drug: Losartan — Losartan is administered orally as pills. It is given preferentially once a day or, if not well tolerated because of hypotension, the total daily dosage is given in two administrations
  Arms: Losartan
Drug: Nebivolol — Nebivolol is administered orally as pills. It is given preferentially once a day in the morning or, if not well tolerated because of hypotension, the total daily dosage is given in two administrations
  Arms: Nebivolol

SUMMARY:
The major clinical problems in patients with Marfan Syndrome (MFS) are aortic root dilation (ARD), dissection and rupture. Although the available treatments (beta-blockers, BBs) improve the evolution of the disease, they do not protect MFS patients from progression of ARD and dissection. A key molecule that negatively influences cell growth, differentiation, survival and death in MFS is TGFb which is antagonised by existing drugs employed in the clinical practice, the Angiotensin II receptor blockers (ARB).

DETAILED DESCRIPTION:
Marfan Syndrome is a rare disease (1:5000)(MIM#154700) caused by mutations of the Fibrillin 1 (FBN1) gene. The major clinical problem is aortic aneurysm with risk of dissection when root diameter is 5 cm.

The investigators designed a clinical trial in which a new generation Beta-Blocker Nebivolol with expected effects on shear stress, heart rate and potential anti-stiffness benefits is compared to Losartan, and Angiotensin receptor blocker anti TGF-beta effects, and to the association of both molecules in patients with Marfan Syndrome. Nebivolol is a patented drug that differs chemically, pharmacologically and therapeutically from all other BBs. Nebivolol shows the highest selectivity for ß1 receptors among the currently available BBs, influences the arterial stiffness through an agonistic effect on ß2-receptors and preserves the arterial compliance. We expect a significantly lower progression of the Aortic Root Dilation in the arm of Nebivolol plus Losartan vs. single drug (primary end-point).The investigators further expect: decrease of arterial stiffness higher in the arm treated with both drugs than in solely Nebivolol or Losartan; a decrease of serum levels of active TGFb in both Losartan arms, a drug & age-dependant variation of the expression of the mutated FBN1 gene. As for other end-points, the potential results are the improvement of valve function, hard events & delay of surgical timing for the aortic root. The enrolment period will last 12 months, while the overall follow-up period will be of 4 years. An interim analysis for the primary outcome is programmed at month 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MFS: Ghent criteria and genetically proven defect of the FBN1 gene
* Age: 12 months to 55 years
* BSA-adjusted aortic z score = or >2 measured at the level of the sinuses of Valsalva at baseline according to Roman's method, or absolute aortic root diameter >38mm for females and >40 mm for males

Exclusion Criteria:

* Prior aortic surgery and/or dissection
* Aortic root diameter at the level of the sinuses of Valsalva 5 cm
* Planned aortic surgery within 6 months of enrollment for a rate of ARD progression>5 mm/year even in pts with ARD less than 5 cm
* Clinical or molecular diagnosis of non-MFS connective tissue diseases sharing some features with MFS (Shprintzen-Goldberg syndrome or Loeys-Dietz syndromes)
* Un-renounceable therapeutic (systemic hypertension, arrhythmia, ventricular dysfunction, valve regurgitation) use of drugs such as ACE inhibitors, BBs, or calcium-channel blockers
* Known side-effects while taking an ARB or a BB
* Intolerance to ARB that resulted in termination of therapy
* Intolerance to BB that resulted in termination of therapy
* Renal dysfunction (creatinine level more than upper limit of age-related normal values)
* Diabetes mellitus
* Pregnancy or planned pregnancy within 48 months of enrollment
* Technical limitations for the imaging studies including poor acoustic windows with limits the accurate measurement of aortic root
* Asthma.

Ages: 12 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 291 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
BSA and age-adjusted aortic root diameter (sinuses of Valsalva) | every 12 months

SECONDARY OUTCOMES:
The pharmacokinetics of the two drugs by age and dosages | every 12 months
Comparative evaluation of the serum levels of total and active TGFb | every 12 months
Quantitative assessment of the expression of the mutated gene (FBN1, both 5' and 3') | every 12 months
Pharmacogenetic bases of drug responsiveness (Losartan: CYP2C9 gene) (Nebivolol: CYP2D6 gene) | every 12 months
Aortic valve regurgitation severity | every 12 months
Left ventricular end-diastolic diameter | every 12 months
Left ventricular ejection fraction | every 12 months
Spirometric lung volumes and flows | every 12 months
QoL evaluation basing on SF-36 questionnaire | every 12 months
Arterial stiffness (carotids) | every 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa Arbustini, MD,FESC,FACC, Principal Investigator — IRCCS Foundation San Matteo Hospital, Pavia; Luigi Tavazzi, MD,FESC,FACC, Study Chair — IRCCS Foundation San Matteo Hospital, Pavia
Locations (1):
- IRCCS Foundation San Matteo Hospital, Pavia, Italy

REFERENCES:
- [Background] Munger JS, Harpel JG, Gleizes PE, Mazzieri R, Nunes I, Rifkin DB. Latent transforming growth factor-beta: structural features and mechanisms of activation. Kidney Int. 1997 May;51(5):1376-82. doi: 10.1038/ki.1997.188. PMID 9150447
- [Background] Hao J, Wang B, Jones SC, Jassal DS, Dixon IM. Interaction between angiotensin II and Smad proteins in fibroblasts in failing heart and in vitro. Am J Physiol Heart Circ Physiol. 2000 Dec;279(6):H3020-30. doi: 10.1152/ajpheart.2000.279.6.H3020. PMID 11087260
- [Background] Border WA, Noble NA. Interactions of transforming growth factor-beta and angiotensin II in renal fibrosis. Hypertension. 1998 Jan;31(1 Pt 2):181-8. doi: 10.1161/01.hyp.31.1.181. PMID 9453300
- [Background] Lim DS, Lutucuta S, Bachireddy P, Youker K, Evans A, Entman M, Roberts R, Marian AJ. Angiotensin II blockade reverses myocardial fibrosis in a transgenic mouse model of human hypertrophic cardiomyopathy. Circulation. 2001 Feb 13;103(6):789-91. doi: 10.1161/01.cir.103.6.789. PMID 11171784
- [Background] Pauwels PJ, Gommeren W, Van Lommen G, Janssen PA, Leysen JE. The receptor binding profile of the new antihypertensive agent nebivolol and its stereoisomers compared with various beta-adrenergic blockers. Mol Pharmacol. 1988 Dec;34(6):843-51. PMID 2462161
- [Background] Ignarro LJ. Experimental evidences of nitric oxide-dependent vasodilatory activity of nebivolol, a third-generation beta-blocker. Blood Press Suppl. 2004 Oct;1:2-16. PMID 15587107
- [Background] McEniery CM, Schmitt M, Qasem A, Webb DJ, Avolio AP, Wilkinson IB, Cockcroft JR. Nebivolol increases arterial distensibility in vivo. Hypertension. 2004 Sep;44(3):305-10. doi: 10.1161/01.HYP.0000137983.45556.6e. Epub 2004 Jul 19. PMID 15262912
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Van Bortel LM, Bulpitt CJ, Fici F. Quality of life and antihypertensive effect with nebivolol and losartan. Am J Hypertens. 2005 Aug;18(8):1060-6. doi: 10.1016/j.amjhyper.2005.03.733. PMID 16296572
- [Background] Mangrella M, Rossi F, Fici F, Rossi F. Pharmacology of nebivolol. Pharmacol Res. 1998 Dec;38(6):419-31. doi: 10.1006/phrs.1998.0387. PMID 9990650
- [Background] Roman MJ, Devereux RB, Kramer-Fox R, O'Loughlin J. Two-dimensional echocardiographic aortic root dimensions in normal children and adults. Am J Cardiol. 1989 Sep 1;64(8):507-12. doi: 10.1016/0002-9149(89)90430-x. PMID 2773795
- [Result] Habashi JP, Judge DP, Holm TM, Cohn RD, Loeys BL, Cooper TK, Myers L, Klein EC, Liu G, Calvi C, Podowski M, Neptune ER, Halushka MK, Bedja D, Gabrielson K, Rifkin DB, Carta L, Ramirez F, Huso DL, Dietz HC. Losartan, an AT1 antagonist, prevents aortic aneurysm in a mouse model of Marfan syndrome. Science. 2006 Apr 7;312(5770):117-21. doi: 10.1126/science.1124287. PMID 16601194
- [Result] Selamet Tierney ES, Feingold B, Printz BF, Park SC, Graham D, Kleinman CS, Mahnke CB, Timchak DM, Neches WH, Gersony WM. Beta-blocker therapy does not alter the rate of aortic root dilation in pediatric patients with Marfan syndrome. J Pediatr. 2007 Jan;150(1):77-82. doi: 10.1016/j.jpeds.2006.09.003. PMID 17188619
- [Result] Ahimastos AA, Aggarwal A, D'Orsa KM, Formosa MF, White AJ, Savarirayan R, Dart AM, Kingwell BA. Effect of perindopril on large artery stiffness and aortic root diameter in patients with Marfan syndrome: a randomized controlled trial. JAMA. 2007 Oct 3;298(13):1539-47. doi: 10.1001/jama.298.13.1539. PMID 17911499 (Retraction: PMID 26594834 JAMA. 2015 Dec 22-29;314(24):2692-3)
- [Derived] Gambarin FI, Favalli V, Serio A, Regazzi M, Pasotti M, Klersy C, Dore R, Mannarino S, Vigano M, Odero A, Amato S, Tavazzi L, Arbustini E. Rationale and design of a trial evaluating the effects of losartan vs. nebivolol vs. the association of both on the progression of aortic root dilation in Marfan syndrome with FBN1 gene mutations. J Cardiovasc Med (Hagerstown). 2009 Apr;10(4):354-62. doi: 10.2459/JCM.0b013e3283232a45. PMID 19430350
- See also: home page of the Polyspecialistic Group for Marfan Syndrome diagnosis and management — http://www.marfansyndrome.eu